CLINICAL TRIAL: NCT05879016
Title: Comparison of the Efficiency of Three Different Taping Methods in Individuals With Myofascial Pain Syndrome With Trigger Point in the Trapezius
Brief Title: Different Taping Methods in Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kubra Koce (Other)
Responsible Party: Sponsor-Investigator, Kubra Koce, Lecturer, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-38
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Myofascial Pain Syndrome; Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Functional Correction Technique
  Interventions: Other: Functional Correction Technique
- Group 2 (Experimental): Fascia Correction Technique
  Interventions: Other: Fascia Correction Technique
- Group 3 (Experimental): Star Taping Technique
  Interventions: Other: Star Taping Technique
- Group 4 (Sham Comparator): I taping technique without tension
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Other: Functional Correction Technique — A single I strip will be used for this technique. Taping will be done by applying moderate (25-35%) degree of stretching to the middle 1/3 of the tape, with the stretched area centered on the trigger point. The ends of the tape will be adhered without stretching.
  Arms: Group 1
Other: Fascia Correction Technique — Y tape will be applied to prevent fascia adhesions. In the Y tape application, first the tail strips of the Y will be adhered with maximum tension so that the muscle fiber is transverse. Then it will be glued so that its base is in front of the pain point. No tension will be applied to the ends of the tape. The application will be applied when the patient is in a resting position and his joints are in a tense position.
  Arms: Group 2
Other: Star Taping Technique — 4 I tapes of the same length between 15 cm and 20 cm will be glued on top of each other. After the first I tape is adhered, the 2nd I tape will be adhered at 90 degrees, then the 3rd and 4th I tapes will be adhered at 45 degrees to obtain a star appearance. There will be no tension at the ends of the tapes
  Arms: Group 3
Other: Sham Comparator — I shape tape will be adhered for sham purpose without applying any tension.
  Arms: Group 4

SUMMARY:
Myofascial pain syndrome is a musculoskeletal pain condition that originates from localized, tight areas of skeletal muscle and fascia, called trigger points. Myofascial pain syndrome is the most common cause of musculoskeletal pain and its prevalence in the community is reported to be 12-55%. Patients with myofascial pain syndrome have pain, stiffness, tenderness, burning, and squeezing sensations in the muscles. In treating myofascial pain syndrome, trigger points should be inactivated and normal body mechanics should be corrected as much as possible. Treatment of the trigger point may be the main goal of a physiotherapy rehabilitation program as it can rapidly reduce acute pain. The goal is to control pain, restore limited ROM, and return the muscle to its optimal length and position. One of the treatment methods applied in MAS is kinesio taping. Kinesio Taping is a non-invasive, painless and less time-consuming method with fewer side effects, widely used as a therapeutic tool in various prevention and rehabilitation protocols. It differs from other rigid tapes because it can stretch significantly (130-140% of its original length), reducing mechanical movement limitations and mimicking skin thickness and elasticity. It has been found to be effective in reducing pain and muscle spasm, increasing range of motion, improving local blood and lymph circulation, reducing edema, strengthening weakened muscles, and controlling joint instability and postural alignment.

Kinesiological tapes can be applied with different shapes and techniques according to the shape and size of the application area and the purpose of the application. Application techniques can be listed as muscle techniques, functional correlation techniques, fascia correlation techniques, star techniques (circulation / lymphatic correction technique), ligament/tendon correction (ligament) technique, mechanical correction techniques, and neural techniques. Functional correlation technique, which is one of the techniques the investigators will prefer in our study, is just above the area of pain, it lifts the skin, fascia, and soft tissue thanks to the elastic properties of the band, thereby reducing the pressure under the application area, reducing the irritation in the chemical receptors and nociceptors, reducing the lymphatic circulation. It is claimed that it increases blood circulation and helps to remove exudate more effectively, and as a result, it helps to reduce pain. The fascia correlation technique, which is the other technique the investigators would prefer to use in our study, is used to bring the fascial tissue to the desired position. The main goal is to reduce tension and adhesions by making vibration (oscillation) movement between the fascia layers. Another technique the investigators will use in our study is the star technique. This technique is aimed at reducing the pressure on the lymphatic vessels and creating a gap that allows circulation in the tissue. Fan-cut tape is often used. Our study aims to compare the effects of 3 different taping techniques (correction, fascia correction, and star technique) in individuals with Myofascial Pain Syndrome with a trigger point in the trapezius muscle.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-30
* Being diagnosed with myofascial pain syndrome
* Pain in the upper trapezius area
* Detection of a taut band in the upper trapezius region on examination
* Presence of at least one active trigger point within the taut band in the upper trapezius -region on examination
* The pain caused by the compression of the trigger point is the pain that the patient complains about
* Having signed the informed consent form

Exclusion Criteria:

* Those who have had major surgery or trauma related to the musculoskeletal system, especially the spine and upper extremities
* Those who have a history of any operation related to the head, neck and shoulder region
* Those with neuromuscular disease
* Those with rheumatic disease in the active period
* Those with systemic diseases (Diabetes, hypothyroidism, infection, malignancy...)
* Those with any pathology related to musculoskeletal disease, especially in the cervical region (cervical discopathy, cervical spondylosis, pathologies related to the shoulder joint and surrounding soft tissues, scoliosis, kyphosis, leg length difference, polio sequelae, developmental hip dysplasia...)
* Those with serious psychological problems (BDI score of 30 and above)
* Those with obesity (BMI≥30 kg/m2)
* Those with tape allergies

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1 week
  The Visual Analogue Scale is a simple, sensitive and reproducible tool that is often used to assess pain severity. Due to its easy application, it has become the most frequently used self-assessment scale in studies on neck pain. It consists of a ten cm long horizontal or vertical line. The starting point of the line represents no pain, and the end represents the most severe pain imaginable. It is stated that the severity of pain increases when the patient goes from the beginning of the line to the end, and the patient is asked to mark the severity of his pain on the line, the point marked by the patient is recorded in cm.
Muscle Strength | 1 week
  With myometer, cervical region flexion, extension, lateral flexion and rotation movements, upper extremity shoulder flexion, abduction, internal and external rotation and elbow flexion angles will be measured bilaterally. Measurements will be repeated 3 times and the average value will be recorded as Newton(N).
Joint Range of Motion | 1 week
  With the universal goniometer, cervical region flexion, extension, lateral flexion and rotation movements, upper extremity shoulder flexion, extension, abduction, adduction, internal and external rotation and elbow flexion and extension angles will be measured bilaterally. Measurements will be repeated 3 times and the average value will be recorded in degrees.
Hand Grip Strength | 1 week
  The maximum isometric contraction strength of the hand and forearm muscles will be measured bilaterally with the hand dynamometer.
Pressure Pain Threshold | 1 week
  The pressure pain threshold that individuals feel will be measured with the Algometer. Algometry is used in many musculoskeletal diseases to evaluate pain and determine therapeutic effects
Number of Active Trigger Points | 1 week
  Trapezius fibers will be evaluated for the number of trigger points by manual palpation.

SECONDARY OUTCOMES:
Nottingham Health Profile | 1 week
  The Nottingham Health Profile was developed in England in 1985 to assess health-related quality of life in individuals and has been translated into many languages. The Nottingham Health Profile is a general quality of life questionnaire that assesses individuals' health problems and the extent to which the problems affect their activities of daily living. The Nottingham Health Profile Questionnaire consists of 38 questions and 6 subtitles. Sub-headings were classified as energy (3 items), social isolation (5 items), pain (8 items), sleep (5 items), physical activity (8 items) and emotional reactions (9 items). The answers to the questions are defined as Yes/No. Each subheading is scored between 0-100. A high total score indicates poor health.
Neck Disability Index | 1 week
  The Neck Disability Index was published in 1991, modified from the Oswestry low back pain disability questionnaire, by Vernon and Mior to evaluate the activities of daily living of patients with neck pain. The Neck Disability Index is the most widely used, translated and the oldest scale in the world to evaluate disability associated with neck pain of non-specific mechanical character. The Neck Disability Index has a total of ten sections. Each section has six possible answers. Each item is scored from 0 (no disability) to 5 (complete disability). The total score ranges from 0 (no disability) to 50 (complete disability) or 0% to 100% in percent terms. With increasing scores, the degree of disability due to neck pain perceived by the patient increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No